CLINICAL TRIAL: NCT01387061
Title: Hepatic Resection for Multiple Hepatocellular Carcinoma on Cirrhosis
Brief Title: Resection for Multiple Hepatocellular Carcinomas (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: multipleHCC
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Hepatocellular Carcinoma; Multiple Tumors; Cirrhosis
Keywords: liver resection; hepatic resection; intraoperative ultrasound
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

ARMS (1):
- hepatic resection (Experimental)
  Interventions: Procedure: hepatic resection

INTERVENTIONS:
Procedure: hepatic resection — surgical resection of the liver for multiple HCC

SUMMARY:
Surgical resection in patients with multiple hepatocellular carcinomas (HCC) remains controversial. The aim of this study was to investigate the outcome of a consecutive cohort of patients resected for multiple HCC, without macrovascular invasion, in order to identify clinically reliable parameters to select patients for surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple HCC without macrovascular invasion on liver cirrhosis

Exclusion Criteria:

* macrovascular invasion;
* normal liver;
* distant or lymphnodes metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2001-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overall survival plus multivariate analysis | 10 years
  The primary endpoint of the study was the overall survival of patients resected for multiple HCC, and the univariate and multivariate analyses of prognostic factors for overall survival.

SECONDARY OUTCOMES:
Disease-free survival | 10 years
  The secondary endpoint was the disease-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Study Chair — University of Milan
Locations (1):
- University of Milan IRCCS Istituto Clinico Humanitas, Rozzano, Milan, MI, Italy